CLINICAL TRIAL: NCT02099032
Title: Influence of Milk Polar Lipids Intake on Lipid Metabolism, Body Composition, Inflammation and Intestinal Microbiota in Menopausal Women
Brief Title: Milk Polar Lipids Consumption, Lipid Metabolism, and Inflammation in Menopausal Women
Acronym: VALOBAB-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013.821
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cardiometabolic Risk
Keywords: nutrition; milk; polar lipids; cardiometabolic risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3g milk polar lipid fortified cheese product (Experimental): Women will have to consume daily 100g of a cheese product instead of usual cheese products during four weeks.
  Interventions: Other: 3g milk polar lipid fortified cheese consumption
- 5 g milk polar lipid fortified cheese product (Experimental): Women will have to consume daily 100g of a cheese product instead of usual cheese products during four weeks.
  Interventions: Other: 5g milk polar lipid fortified cheese consumption
- Unfortified cheese product (Placebo Comparator): Women will have to consume daily 100g of a cheese product instead of usual cheese products during four weeks
  Interventions: Other: Unfortified cheese product consumption

INTERVENTIONS:
Other: 3g milk polar lipid fortified cheese consumption — Women will have to consume daily 100g of a 3g milk polar lipid fortified cheese product instead of usual cheese products during four weeks.
  Arms: 3g milk polar lipid fortified cheese product
Other: 5g milk polar lipid fortified cheese consumption — Women will have to consume daily 100g of a 5 g milk polar lipid fortified cheese product instead of usual cheese products during four weeks.
  Arms: 5 g milk polar lipid fortified cheese product
Other: Unfortified cheese product consumption — Women will have to consume daily 100g of a unfortified cheese product instead of usual cheese products during four weeks
  Arms: Unfortified cheese product

SUMMARY:
Polar lipids have a specific chemical structure: they are an essential component of human cell membranes, play a major role in the nervous system and also influence the metabolic pathways including the cholesterol metabolism.

Polar lipids are used in food-processing industry for their emulsification properties. The most famous emulsifier is soya lecithin but milk also naturally contains natural emulsifiers such as polar lipids.

The purpose of this research is to study plasma cholesterol variation after daily intake of milk polar lipids-fortified cheese products. The volunteers will have to consume 100 g of cheese product during four weeks instead of their usual cheese products.

It is a bi-centric study with a centre in LYON (Centre de Recherche en Nutrition Humaine Rhône-Alpes) and CLERMONT-FERRAND (Centre de Recherche en Nutrition Humaine Auvergne).

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women
* Of less than 75 years old- Body Mass Index of 25 to 35 kg/m2
* Waist circumference greater than 80 cm
* Normal (or not clinically significant) glycemic and lipid parameters

Exclusion Criteria:

* Dairy products allergy or intolerance
* Smokers (more than five cigarettes/day)
* HDL cholesterol greater than 1.5 mmol/L
* Medication that could interfere with lipid metabolism or intestinal microbiota (for example, no antibiotics within the 2 months before the study)
* Hormone replacement treatment for menopause

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Total plasma cholesterol | Day 0 and Day 28
  Total plasma cholesterol will be measured fasting before and after the four weeks of cheese product intake.

SECONDARY OUTCOMES:
Plasma lipids | Day 0 and Day 28
  Plasma lipids will be measured before and after the four weeks of cheese product intake. Fasting and postprandial measurements over 8 hours depending on parameters (time 60-120-180-240-270-300-360-420-480 minutes)
Plasma glucose and insulin | Day 0 and Day 28
  Plasma glucose and insulin will be measured before and after the four weeks of cheese product intake. Fasting and postprandial measurements over 8 hours.
Inflammatory markers | Day 0 and Day 28
  Inflammatory markers will be measured before and after the four weeks of cheese product intake. Fasting and postprandial measurements over 8 hours depending on parameters
Body composition measurement with bioimpedancemetry | Day 0 and Day 28
  Body composition will be measured fasting before and after the four weeks of cheese product intake.
Energy expenditure and substrate oxidation with indirect calorimetry | Day 0 and Day 28
  Energy metabolism will be measured before and after the four weeks of cheese product intake. Fasting and during all the postprandial period (480 minutes)
Intestinal microbiota with molecular approach | before and after the four weeks of cheese product intake
  Stools will be collected at home before and after the four weeks of cheese product intake.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Université d'Auvergne-Laboratoire de Nutrition Humaine, Clermont-Ferrand
  - Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite

REFERENCES:
- [Derived] Le Barz M, Vors C, Combe E, Joumard-Cubizolles L, Lecomte M, Joffre F, Trauchessec M, Pesenti S, Loizon E, Breyton AE, Meugnier E, Bertrand K, Drai J, Robert C, Durand A, Cuerq C, Gaborit P, Leconte N, Bernalier-Donadille A, Cotte E, Laville M, Lambert-Porcheron S, Ouchchane L, Vidal H, Malpuech-Brugere C, Cheillan D, Michalski MC. Milk polar lipids favorably alter circulating and intestinal ceramide and sphingomyelin species in postmenopausal women. JCI Insight. 2021 May 24;6(10):e146161. doi: 10.1172/jci.insight.146161. PMID 33857018
- [Derived] Vors C, Joumard-Cubizolles L, Lecomte M, Combe E, Ouchchane L, Drai J, Raynal K, Joffre F, Meiller L, Le Barz M, Gaborit P, Caille A, Sothier M, Domingues-Faria C, Blot A, Wauquier A, Blond E, Sauvinet V, Gesan-Guiziou G, Bodin JP, Moulin P, Cheillan D, Vidal H, Morio B, Cotte E, Morel-Laporte F, Laville M, Bernalier-Donadille A, Lambert-Porcheron S, Malpuech-Brugere C, Michalski MC. Milk polar lipids reduce lipid cardiovascular risk factors in overweight postmenopausal women: towards a gut sphingomyelin-cholesterol interplay. Gut. 2020 Mar;69(3):487-501. doi: 10.1136/gutjnl-2018-318155. Epub 2019 Jun 12. PMID 31189655
- See also: Related Info — http://www.crnh-rhone-alpes.fr
- See also: Related Info — http://www1.clermont.inra.fr/crnh/